CLINICAL TRIAL: NCT05095259
Title: Metabolic Adaptation to High-frequent Hypoglycaemia in Type 1 Diabetes - the HypoADAPT Study
Brief Title: Metabolic Adaptation to High-frequent Hypoglycaemia in Type 1 Diabetes
Acronym: HypoADAPT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nordsjaellands Hospital (Other)
Collaborators: Danish Research Centre for Magnetic Resonance (Other); University of Copenhagen (Other); Steno Diabetes Center Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: DRCMR7T-06; 2019-001938-34 (EudraCT Number)
Record Dates: First submitted 2021-10-01; First posted 2021-10-27 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-02

CONDITIONS: Type1diabetes
Keywords: Diabetes Complications; Hypoglycemia; Metabolism
MeSH Terms: conditions — Diabetes Complications; Hypoglycemia | interventions — Insulin; Epinephrine; Glucagon; Glucagon-Like Peptide 1; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Intervention Model Description: Experimental Observational Case-Control study. Two groups: One group of type 1 diabetes and one group of healthy controls.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Participants with Type 1 Diabetes Mellitus (Experimental): Participants with Type 1 Diabetes Mellitus
  Interventions: Drug: insulin human; Drug: Epinephrin; Procedure: Muscle biopsy; Procedure: Adipose tissue biopsy; Drug: Glucagon; Device: IPRO 2 Medtronic Minimed; Procedure: 7 Tesla (7T) Magnetic Resonance Imaging; Procedure: Indirect Calorimetry using Jaeger Oxycon Champion; Procedure: Core temperature and thermography using Thermovision SC645; Device: Freestyle Libre 2
- Healthy Controls (Active Comparator): Healthy Controls
  Interventions: Drug: insulin human; Drug: Epinephrin; Procedure: Muscle biopsy; Procedure: Adipose tissue biopsy; Drug: Glucagon; Device: IPRO 2 Medtronic Minimed; Procedure: 7 Tesla (7T) Magnetic Resonance Imaging; Procedure: Indirect Calorimetry using Jaeger Oxycon Champion; Procedure: Core temperature and thermography using Thermovision SC645

INTERVENTIONS:
Drug: insulin human — Hyperinsulinemic glucose clamp studies require that insulin is administered at a steady continuous rate to achieve stable levels of hyperinsulinemia. To reach this, insulin needs to be infused intravenously using a standard intravenous pump system. The insulin dose will be adjusted according to the body surface area, aiming for insulin levels of ~170 mIU/l, which is within the physiological range. Thus, for a subject with a bodyweight of 70 kg, body length of 180 cm and - consequently - a body surface area of 1.936 m2, the required insulin infusion can be calculated as: 1.936 x 60 x 60 ÷ 1000 = 7.0 units per hour
  Other Names: Actrapid
Drug: Epinephrin — Epinephrine are prepared in 100 ml isotone saline solution according to weight and infused in 3 different infusion rates: 10 ng∙kg-1∙min-1, 25 ng∙kg-1∙min-1 and 50 ng∙kg-1∙min-1, for 20 minutes each. After each adrenaline infusion, substrate response will be measured by blood samples of glucose, lactate, free fatty acids, alanine, β-hydroxybutyrate, glycerol and insulin. Furthermore, cardiovascular measurements such as pulse and blood pressure are monitored as well.
  Other Names: Adrenalin
Procedure: Muscle biopsy — With the study subject resting in the supine position, the skin is disinfected on the lateral side of the thigh around 15 cm above the knee, with chlorhexidine alcohol. Then 3-4 mL of local anaesthetic (lidocaine 20 mg/mL) is injected into the skin, subcutaneous tissue and in the upper part of the muscle with a very thin needle. When the anaesthetic effect has set in after a couple of minutes an insertion is made in the skin and the subcutaneous tissue through which the biopsy cannula is inserted into the muscle. A small piece (around 150 mg) of the muscle is collected, which may be experienced as somewhat unpleasant, but will last for a very short while ( ~1-2 seconds). The needle is removed, a sterile Band-Aid is applied, and the study subject can leave the site after termination of the trial. The biopsy may cause some muscular tenderness for 2-3 days corresponding to minor muscular trauma.
Procedure: Adipose tissue biopsy — With the study subject resting in the supine position, the skin is disinfected on one side of the abdomen around 5-10 cm lateral from the umbilicus to the knee, with chlorhexidine alcohol. Then 3-4 mL of local anaesthetic (lidocaine 20 mg/mL) is injected into the skin, subcutaneous tissue and in the upper part of the adipose tissue with a very thin needle. When the anaesthetic effect has set in after a couple of minutes an insertion is made in the skin and the subcutaneous tissue through which the biopsy cannula is inserted into the adipose tissue. A small piece (around 1 gram) of the adipose tissue is collected, which may be experienced as somewhat unpleasant, but will last for a very short while ( ~1-2 seconds). The needle is removed, a sterile Band-Aid is applied, and the study subject can leave the site after termination of the trial. The biopsy may cause some tenderness for 2-3 days corresponding to minor trauma.
Drug: Glucagon — Glucagon is prepared in doses of 10 µg, 25 µg, and 50 µg and intravenously injected with intervals of 2 hours. After each glucagon injection, blood samples will be drawn to measure plasma glucose, glucagon, lactate, free fatty acids, alanine, amino-acids, β-hydroxybutyrate, glycerol and insulin. Furthermore, cardiovascular measurements such as pulse and blood pressure are monitored as well.
  Other Names: GlucaGen
Device: IPRO 2 Medtronic Minimed — All potential subjects will receive a blinded continuous glucose sensor at Visit 1. At the following visits, the continuous glucose monitor (CGM) will be reviewed for hypoglycaemia episodes and replaced at the same time. At Visit 2 a final screening of the inclusion criteria will take place, which involves the CGM data of the first week. A blinded CGM will be installed a week before every visit.
  Other Names: Blinded Continuous Glucose Monitoring
Procedure: 7 Tesla (7T) Magnetic Resonance Imaging — Subjects will undergo a hyperinsulinemic euglycaemic glucose clamp, as mentioned above, in the MRI scanning room. After 30 minutes of stable normoglycaemia, subjects are taken into the MRI scanner (Philips Achieva 7.0 T) where brain, liver, thigh and calf muscle are scanned. After every anatomically different area, the subjects must be taken out of the scanner, while scanning coils are replaced. All subjects are advised to lie still and press the alarm button if necessary.
  Other Names: 7T MRI
Procedure: Indirect Calorimetry using Jaeger Oxycon Champion — Resting metabolic rate will be estimated, after reaching stable plasma glucose level, via a hyperinsulinemic euglycaemic clamp, as mentioned above. This will be done by indirect calorimetry, using a ventilated hood system (Jaeger Oxycon Champion, software version 4.3, Jaeger, Mijnhardt). Subjects are instructed to lie down and rest for a period of 30 minutes. Subjects are also instructed not to move, talk or sleep unless necessary during the period of measurement. The recorded measurement after 5 minutes to 30 minutes will be used for analysis.
Procedure: Core temperature and thermography using Thermovision SC645 — Thermography (Thermovision SC645, FLIR Systems, Wilsonville, OR, USA) is used to determine cutaneous vascular perfusion. Data is analogue-digital converted and sampled at 100 Hz (Powerlab, ADInstruments, Colorado Springs, CO, USA).
Device: Freestyle Libre 2 — All potential subjects will receive a continuous glucose sensor at Visit 1. At the following visits, the CGM will be reviewed for hypoglycaemia episodes and replaced at the same time. At Visit 2 a final screening of the inclusion criteria will take place, which involves the CGM data of the first week. A CGM will be installed a week before every visit.
  Other Names: Intermittently scanned continuous glucose monitor
  Arms: Participants with Type 1 Diabetes Mellitus

SUMMARY:
An experimental mechanistic study. The overall objective is to gain new knowledge about mechanisms involved in adaptation to recurrent hypoglycaemia in diabetes by investigating patients with type 1 diabetes and healthy controls. The knowledge to be obtained may feed into experimental hypoglycaemic clamp studies to further elucidate the effect of the adaptations during acute hypoglycaemia. Ultimately, it may lead to intervention studies aiming at the maintenance of functional capability during hypoglycaemia in patients with type 1 diabetes to reduce their risk of severe hypoglycaemia.

DETAILED DESCRIPTION:
Study rationale The risk of severe hypoglycaemia is a major daily concern for people with diabetes treated with insulin. Severe hypoglycaemia is the main barrier in achieving the recommended glycaemic targets and may indirectly be the main driver for late diabetic complications and related morbidity, mortality and health care costs. In people with diabetes, recurrent exposure to insulin-induced mild hypoglycaemia leads to significant adaptive physiologic responses. While the metabolism of the brain and hormonal responses to hypoglycaemia have been studied extensively, this study will as the first, systematically investigate the chronic adaptation of peripheral metabolism to recurrent hypoglycaemia in diabetes. Knowledge about such responses can lead to interventions that attenuate the devastating effects of acute hypoglycaemia induced by insulin in people with diabetes. Thereby, the risk of developing severe hypoglycaemia can be reduced which ultimately will improve long-term diabetes outcomes and reduce health care costs.

Hypothesis Patients with type 1 diabetes that are exposed to high-frequent recurrent hypoglycaemia will adapt their metabolism in a way, which supports the preservation of brain fuelling.

Objectives

Primary objective The overall objective is to gain new knowledge about mechanisms involved in adaptation to recurrent hypoglycaemia in diabetes by investigating patients with type 1 diabetes and healthy controls. The knowledge to be obtained may feed into experimental hypoglycaemic clamp studies to further elucidate the effect of the adaptations during acute hypoglycaemia. Ultimately, it can lead to intervention studies aiming at the maintenance of functional capability during hypoglycaemia in patients with type 1 diabetes to reduce their risk of severe hypoglycaemia.

Secondary objectives

* To study the metabolic consequences of recurrent hypoglycaemia in the brain, liver, muscle and adipose tissues
* To study the consequences of recurrent hypoglycaemia on resting metabolic rest
* To study the consequences of recurrent hypoglycaemia on glucagon and adrenaline sensitivity
* To study the consequences of recurrent hypoglycaemia on epigenetic profiles
* To study the consequences of recurrent hypoglycaemia on oxidative stress
* To study the psychological factors associated with recurrent hypoglycaemia

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide written informed consent
2. Male or female aged 18-70 years
3. Must be able to speak and read Danish
4. Type 1 diabetes patients or healthy individuals (control goup)
5. A documented clinically relevant history of type 1 diabetes
6. In insulin treatment regimen
7. The subject must be willing and able to comply with trial protocol

Exclusion Criteria:

1. History of severe psychological condition
2. History of severe heart disease
3. History of epilepsy, former apoplexies and dementia
4. History of muscle diseases
5. History of liver disease
6. History of malignancy unless a disease-free period exceeding 5 years
7. Implants not compatible for MRI scans
8. History of alcohol or drug abuse
9. Pregnant or lactating woman

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-12-16 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Metabolite- and lipid profiling | 5 minutes
  Metabolite- and lipid profiling of blood samples using metabolomics profiling platforms during euglycaemia
Brain lactate concentration | 20 minutes
  Brain lactate concentration using non-invasive magnetic resonance (MR) spectroscopy during euglycaemia
Brain adenosine triphosphate (ATP) concentration | 20 minutes
  Brain ATP concentration using non-invasive MR spectroscopy during euglycaemia
Glycogen in muscle and adipose tissue | 5 minutes
  Glycogen in muscle and adipose tissue biopsies during euglycaemia
Non-specific proteins in muscle and adipose tissue | 5 minutes
  Non-specific proteins in muscle and adipose tissue biopsies during euglycaemia
Glycogen concentration | 40 minutes
  Glycogen in liver and muscle tissue using non-invasive MR spectroscopy during euglycaemia.

SECONDARY OUTCOMES:
Estimated glucose production during glucagon stimulation | Every 5 minutes up to 5 hours
  Area under the curve (AUC) for plasma glucose during glucagon injections. Plasma glucose measurement
Estimated glucose production during epinephrine stimulation | Every 5 minutes up to 90 minutes
  Area under the curve (AUC) for plasma glucose during epinephrine infusion. Plasma glucose measurement
Indirect calorimetry | 60 minutes
  Estimating resting metabolic rate, before and during hyperinsulinemic-hypoglycemic clamp
Thermography | 5 minutes
  Estimating skin temperature, before and during hyperinsulinemic-hypoglycemic clamp
Plasma lactate during glucagon injections. | Every 40 minutes up to 5 hours
  Plasma lactate during glucagon injections.
Plasma free fatty acids during glucagon injections. | Every 40 minutes up to 5 hours
  Plasma free fatty acids during glucagon injections.
Plasma glycerol during glucagon injections. | Every 40 minutes up to 5 hours
  Plasma glycerol during glucagon injections.
Plasma alanine during glucagon injections. | Every 40 minutes up to 5 hours
  Plasma alanine during glucagon injections.
Plasma β-hydroxybutyrate during glucagon injections. | Every 40 minutes up to 5 hours
  Plasma β-hydroxybutyrate during glucagon injections.
Plasma insulin during glucagon injections. | Every 40 minutes up to 5 hours
  Plasma insulin during glucagon injections.
Plasma glucagon during glucagon injections. | Every 40 minutes up to 5 hours
  Plasma glucagon during glucagon injections.
Plasma metabolomics during glucagon injections. | Every 40 minutes up to 5 hours
  Plasma metabolomics during glucagon injections.
Plasma lactate during epinephrine infusion | Every 20 minutes up to 90 minutes
  Plasma lactate during epinephrine infusion
Plasma free fatty acids during epinephrine infusion | Every 20 minutes up to 90 minutes
  Plasma free fatty acids during epinephrine infusion
Plasma glycerol during epinephrine infusion | Every 20 minutes up to 90 minutes
  Plasma glycerol during epinephrine infusion
Plasma alanine during epinephrine infusion | Every 20 minutes up to 90 minutes
  Plasma alanine during epinephrine infusion
Plasma β-hydroxybutyrate during epinephrine infusion | Every 20 minutes up to 90 minutes
  Plasma β-hydroxybutyrate during epinephrine infusion
Plasma insulin during epinephrine infusion | Every 20 minutes up to 90 minutes
  Plasma insulin during epinephrine infusion
Plasma glucagon during epinephrine infusion | Every 20 minutes up to 90 minutes
  Plasma glucagon during epinephrine infusion
Plasma epinephrine during epinephrine infusion | Every 20 minutes up to 90 minutes
  Plasma catecholamines during epinephrine infusion
Plasma norepinephrine during epinephrine infusion | Every 20 minutes up to 90 minutes
  Plasma catecholamines during epinephrine infusion
Plasma metabolomics during epinephrine infusion | Every 20 minutes up to 90 minutes
  Plasma metabolomics during epinephrine infusion
Personality traits using the psychometry questionnaire Type D Scale-14 (DS-14) | 30 minutes
  Personality traits using the psychometry questionnaire DS-14, score between 0-28, the higher, the more likely they have type D personality
Personality traits using the psychometry questionnaire Toronto Alexithymia Scale (TAS-20) | 30 minutes
  Personality traits using the psychometry questionnaire TAS-20, score 20-100, the higher score the more likely they are alexithymia
Diabetes and hypoglycaemia status using psychometry questionnaire Hypoglycemia Fear Survey - Worry (HFS-W) | 30 minutes
  Diabetes and hypoglycaemia status using psychometry questionnaire HFS-W, score 0-72, the higher score the higher fear for hypoglycemia
Diabetes and hypoglycaemia status using psychometry questionnaire Hypoglycemia Attitudes and Behavior Scale (HABS) | 30 minutes
  Diabetes and hypoglycaemia status using psychometry questionnaire HABS, score from 14-45, higher score more fear of hypoglycemia
Diabetes and hypoglycaemia status using psychometry questionnaire Problem Areas in Diabetes (PAID) | 30 minutes
  Diabetes and hypoglycaemia status using psychometry questionnaire PAID, 0-80, the higher score, the more problems with diabetes
Food consumption | 30 minutes
  Using Food Frequency Questionnaire to analyze food consumption
Hypoglycemia awareness status | 10 minutes
  Using hypoglycemia awareness status questionnaire
  , 0-7, higher score indicate hypoglycemia unawareness

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik Pedersen-Bjergaard, MD,PhD,Prof, Principal Investigator — Nordsjaellands Hospital
Locations (2):
- Denmark (2):
  - Steno Diabetes Center Copenhagen, Gentofte Municipality
  - Nordsjaellands Hospital, Hillerød

REFERENCES:
- [Derived] She R, Suvitaival T, Andersen HU, Hommel E, Norgaard K, Wojtaszewski JFP, Legido-Quigley C, Pedersen-Bjergaard U. Metabolic effect of adrenaline infusion in people with type 1 diabetes and healthy individuals. Diabetologia. 2024 Jun;67(6):1095-1106. doi: 10.1007/s00125-024-06116-5. Epub 2024 Mar 1. PMID 38427076